CLINICAL TRIAL: NCT01383551
Title: "Becoming Parents": A Hospital-community Partnership to Enhance Transition to Parenthood
Brief Title: "Becoming Parents": A Hospital-community Partnership
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Princess Margaret Hospital, Hong Kong (Other Government); Kwong Wah Hospital (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, TIWARI, Agnes, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 11-163
Record Dates: First submitted 2011-05-30; First posted 2011-06-28 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Expectant Couples
Keywords: Depression; Marital relationship; Parental competence
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Becoming Parents" intervention (Experimental): A "Becoming Parents" Programme consists of: (i) 3 antenatal workshops conducted over a period of 10-14 weeks in prenatal period; and (ii) support provided by trained volunteers for up to 3 months post-delivery; in addition to the usual prenatal education.
  Interventions: Behavioral: "Becoming Parents" intervention
- Usual prenatal education (No Intervention): Attend usual prenatal classes which will be provided by the midwives in the hospital.

INTERVENTIONS:
Behavioral: "Becoming Parents" intervention — A "Becoming Parents" programme consists of: (i) 3 antenatal workshops conducted over a period of 10-14 weeks in prenatal period; and (ii) support provided by trained volunteers for up to 3 months post-delivery; in addition to the usual prenatal education.
  Arms: "Becoming Parents" intervention

SUMMARY:
The proposed of this study is to determine if an intervention, known as the "Becoming Parents" programme, is more effective in improving the mental health, marital relationship and parental competence of expectant couples in a Chinese community.

DETAILED DESCRIPTION:
Transition to parenthood is potentially a stressful life event for many new parents, which, if not properly managed, could have adverse effects on their mental health, marital satisfaction, and parent-child relationships. The proposed programme, "Becoming Parents", aims to turn the challenges of the transition into opportunities of learning and support for these parents. Building on our experience of instituting a pioneering programme to support new fathers prenatally, "Becoming Parents" has an extra component of support for new parents in the postnatal period using trained volunteers from the community networks. Through "Becoming Parents", seamless antenatal-postnatal care based on a hospital-community partnership will be provided to 125 expectant couples in a target community which is known for its high risks for postnatal depression, child abuse and intimate partner violence. In addition to addressing the health promotional needs of the target community, "Becoming Parents" will also illustrate how a community's capacity for health promotion can be maximized through the collaboration of healthcare providers and network of community partners in helping couples function more optimally during their transition to parenthood.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Expectant couples with the pregnant women attending antenatal clinic in Princess Margaret Hospital before 20 weeks of gestation.

Exclusion Criteria:

1. Expected couples who are unable to communicate in Cantonese, Putonghua or English.
2. Multiple pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Depressive Symptoms at 3 months postpartum | Baseline and 3 months postpartum
  The Edinburgh Postnatal Depression Scale is used to measure women's distressed mood or dysphoria at baseline and also at 3 months postpartum

SECONDARY OUTCOMES:
Change from Baseline in Parental Competence at 3 months postpartum | Baseline and 3 months postpartum
  The Parental Sense of Competence Scale is used to measure parenting efficacy and satisfaction at baseline and also at 3 months postpartum
Change from Baseline in Marital Satisfaction at 3 months postpartum | Baseline and 3 months postpartum
  The Dyadic Adjustment Scale is used to measure couples' consensus, cohesion, satisfaction and affection expression at baseline and also at 3 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Tiwari, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Princess Margaret Hospital, New Territories, Hong Kong

REFERENCES:
- [Background] Aston ML. Learning to be a normal mother: empowerment and pedagogy in postpartum classes. Public Health Nurs. 2002 Jul-Aug;19(4):284-93. doi: 10.1046/j.1525-1446.2002.19408.x. PMID 12071902
- [Background] Doherty WJ, Erickson MF, LaRossa R. An intervention to increase father involvement and skills with infants during the transition to parenthood. J Fam Psychol. 2006 Sep;20(3):438-47. doi: 10.1037/0893-3200.20.3.438. PMID 16938002
- [Background] Walther VN. Postpartum depression: a review for perinatal social workers. Soc Work Health Care. 1997;24(3-4):99-111. doi: 10.1300/J010v24n03_08. PMID 9127907
- [Background] Draper J. Men's passage to fatherhood: an analysis of the contemporary relevance of transition theory. Nurs Inq. 2003 Mar;10(1):66-77. doi: 10.1046/j.1440-1800.2003.00157.x. PMID 12622806
- [Background] Belsky, J., & Pensky, E. (1998). Marital change across the transition to parenthood. Marriage and Family Review, 12, (3-4), 133-156.
- [Background] Krishnakmuar, A., & Buehler, C. (2000). Inter-parental conflict and parenting behaviours: A meta-analytic review. Family Relations, 49, 25-44.
- [Background] Cowan, C., & Cowan P. (1995). Interventions to ease the transition to parenthood: Why they are needed and what they can do. Family Relations, 44, 412-414.
- [Background] Markman, H., & Hahlweg, K. (1993). The prediction and prevention of marital distress: an international perspective. Clinical Psychology Review, 13, 29-43.
- [Background] Minsky, R., Garfinkel, I., & Neprmnyaschy, L. (2005). In-hospital paternity establishment and father involvement in fragile families. Journal of Marriage and the Family, 67(3), 611-626.
- [Background] Gottman, J.M., Shapiro, A.F. Parthemer, J. (2004). Bringing Baby Home: A workshop for new and expectant parents. International Journal of Childbirth Education, 19(3), 28-30.
- [Background] Early, R. (2001). Men as consumers of maternity services: a contradiction in terms. International Journal of Consumer Studies, 25, 160-167.
- [Background] Tiwari, A. Leung, W.C., Yuen, K.H., & Wong, J. (2010). Positive fathering: A programme to enhance the mental health and marital relationship of expectant couples. A progress report for a HCPF-funded project submitted to Research Fund Secretariat, Health Care and Promotion Fund Committee on June 29, 2010.